CLINICAL TRIAL: NCT01501565
Title: Ultrasound-guided Analgesic Transverse Abdominal Plain Blockade in the Multimodal Pain Management for Laparoscopic Urological Surgery. Analgesic Efficacy Assessment.
Brief Title: Analgesic Efficacy of Ultrasound-guided Transverse-abdominal Plain Blockade in Urological Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacio Puigvert (Other)
Responsible Party: Principal Investigator, Juan Francisco Mayoral Farre, Principal Investigator, Fundacio Puigvert
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FP2011/01; 2011-003219-53 (EudraCT Number)
Record Dates: First submitted 2011-12-22; First posted 2011-12-29 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Transverse abdominal blockade; Efficacy; Safety; Urology
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard analgesic therapy: iv Metamizol 2 g q8h
- TAP (Experimental): Transverse abdominal plain (TAP) blockade with local anesthetic: Bupivacaine chlorhydrate 0.25% adjusted by weight and type of surgery. Maximum dose: 150 mg of bupivacaine.
  Two approaches are done: 1)Posterior TAP: the needle insertion point is cephalad to the iliac crest, behind the midaxillary line. The needle is inserted under ultrasound guidance in plane. Local anesthetics is deposited between the internal oblique and transversus abdominis muscles, 2)Subcostal TAP: the needle is inserted ultrasound guided perpendicularly to abdominal wall, directed parallel to the costal margin but oblique to the sagittal plane. Local anesthestic is deposited between transversus abdominis and the rectus abdominis muscles.
  Interventions: Procedure: Postoperative transverse abdominal plain (TAP) blockade

INTERVENTIONS:
Procedure: Postoperative transverse abdominal plain (TAP) blockade — Bupivacaine 0.25%. Maximum 150 mg. A maximum of 75 mg bupivacaine is administered in each side (posterior and subcostal TAP) in a single puncture.
  Other Names: Buivacaine: Inibsicain (R) 0.25% (INIBSA, S.A.)
  Arms: TAP

SUMMARY:
The purpose of this study is to compare pain level (according to numerical score)at 4, 8, 12 and 24 postoperative hours between patients under transverse abdominal plain blockade (TAP) and patients under conventional analgesia. Also the opioid consumption is assessed.

ELIGIBILITY:
Inclusion Criteria:

* > 18 yrs.
* Patients undergo laparoscopic urologic surgery
* Physical status ASA < 3
* Surgical procedure without complications
* Signed informed consent

Exclusion Criteria:

* Allergy to bupivacaine chlorhydrate
* Patients with chronic pain treatment
* Alcoholism
* Decompensated hepatic disease
* Coagulation disorders
* BMI > 35
* Patient involved in another clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2011-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pain level | Change in pain from admittance to 24 hours postoperatively
  Pain is assessed by numerical scale (0 to 10) where 0 is no pain and 10 is the most intense pain possible. Pain will be assessed at 4, 6 , 8, 12 and 24 hours.

SECONDARY OUTCOMES:
Analgesic consumption as a rescue therapy | within 24 postoperative hours
  Analgesic consumption: morphine in miligrams.
Incidence of postoperative nausea and vomiting (PONV) related to therapy | within 24 postoperative hours
  Assessment of PONV incidence and antiemetic drugs consumption.
Incidence of urethral/bladder spasm | within 24 postoperative hours
  Pain due to bladder catheter.
Assessment of oral intake tolerance | within 24 postoperative hours
  Assessment at 6 postoperative hours for liquids, and solid food at 24 postoperative hours.
Patient satisfaction | within 24 postoperative hours
  Assessed by ordinal scale: Very pleased/Pleased/little pleased/little unpleased/unpleased/very unpleased

CONTACTS AND LOCATIONS:
Overall Officials: Juan Francisco Mayoral, MD, Principal Investigator — Fundació Puigvert (IUNA)
Locations (1):
- Fundació Puigvert, Barcelona, Barcelona, Spain